CLINICAL TRIAL: NCT00874276
Title: Pharmacotoxicology of Trichloroethylene Metabolites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 14617-CP-004; NCT00874705 (obsolete NCT alias)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Results first posted 2013-06-20 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2013-03

CONDITIONS: Congenital Lactic Acidosis
Keywords: DCA; Dichloroacetate; Trichloroacetate
MeSH Terms: interventions — Dichloroacetic Acid; Genotype; Genetic Markers; Haplotypes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No EGT Allele, slow metabolizers for DCA (Experimental): Individuals were genotyped at the beginning of the study and their haplotypes were defined. Dichloroacetate 2.5.ug/kg (non-clinical dose) will be administered for five days in the clinical research center. On day 5 with the dose of DCA a pharmacokinetics test will be performed for 24 hours. 30 days later the individuals will return to the clinic and receive Dichloroacetate 25mg/kg (clinical dose) for five days. On day 1 and day 5 Pharmacokinetics will be performed to determine the relationship between DCA metabolism and haplotype.
  Interventions: Drug: Dichloroacetate (DCA); Genetic: Genetic Marker on Chromosome 14q24.3
- 1+ EGT Allele, fast metabolizers for DCA (Experimental): Individuals were genotyped at the beginning of the study and their haplotypes were defined. Dichloroacetate 2.5.ug/kg (non-clinical dose) will be administered for five days in the clinical research center. On day 5 with the dose of DCA a pharmacokinetics test will be performed for 24 hours. 30 days later the individuals will return to the clinic and receive Dichloroacetate 25mg/kg (clinical dose) for five days. On day 1 and day 5 Pharmacokinetics will be performed to determine the relationship between DCA metabolism and haplotype.
  Interventions: Drug: Dichloroacetate (DCA); Genetic: Genetic Marker on Chromosome 14q24.3

INTERVENTIONS:
Drug: Dichloroacetate (DCA) — Dichloroacetate 2.5.ug/kg will be administered for five days in the clinical research center. On day 5 with the dose of DCA a pharmacokinetics test will be performed for 24 hours. 30 days later the individuals will return to the clinic and receive Dichloroacetate 25mg/kg (clinical dose) for five days. On day 1 and day 5 Pharmacokinetics will be performed to determine the relationship between DCA metabolism and haplotype.
  Other Names: genotype
Genetic: Genetic Marker on Chromosome 14q24.3 — Individuals were genotyped at the beginning of the study and their haplotypes were defined. The study is looking at individuals with genetic markers on Chromosome 14q24.3 to determine if there will be a difference in how the DCA will be metabolized.
  Other Names: Genetic Marker; Haplotypes

SUMMARY:
To establish the relationship between human MAAI haplotype and DCA and tyrosine metabolism. This aim test the postulates that MAAI haplotype determines, and thus can predict,1) dose-dependent DCA kinetics and biotransformation.

DETAILED DESCRIPTION:
The arms of the study involves determining the haplotype of individuals enrolled. Then participants were divided into two groups based on their genotype. The groups include a genotype with an EGT alle and a group of genotype without an EGT alle. All subjects first took a low dose of DCA 2.5ug/kg for 5 days then wait 30 days and take a therapeutic dose of DCA 25mg/kg for 5 days On the first day and on the 5th day of taking DCA kinetics were be done. A total of 16 blood samples were obtained through an intravenous catheter. Urine collection will also occur.

Population pharmacogenetic analysis of MAI allelic frequencies and the GC or LC-MS/MS techniques for blood or urinary metabolites were used in this investigation. Pharmacokinetic data was used to determine metabolism rate of DCA for each allele

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Pregnancy
* Other medications
* Psychiatric illness on meds
* Abnormal labs

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2009-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter W Stacpoole, PhD, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Shands Hospital, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from a list of individuals who had already been genotyped. Subjects were called on the telephone to see if they wanted to participate in this study.
Pre-assignment Details: 21 subjects were consented to the study; however, 7 were excluded before being assigned to a group for the following reasons: works at night, on contraindicated medication, history of mitral valve prolapse, obesity, started smoking, and elevated liver enzymes.
Groups:
- Lack Any EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3; 1+ EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3: Both dichloroacetate 2.5ug and 25mg per kg per day and is administered for five days. (Biologic randomization)
  Dichloroacetate 2.5ug/kg (Environmental) and 25mg/kg (clinical) are administered daily for 5 days in all subjects. Subjects are admitted to the clinical research center for 6 nights. The first day subjects are administer 2.5ug/kg/day. Frequent blood samples are collected over a 24 hour period. On days 2, 3, 4 the subjects receive a dose of DCA each day. On day 5 they receive a dose of DCA and pharmacokinetics are done for 24 hours then subjects are discharged.
Period: Overall Study
Arm/Group | Lack Any EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3 | 1+ EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3
Started | 6 | 8
Completed | 5 | 7
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Lack Any EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3; 1+ EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3: This study is a biological randomization for dichloroacetate pharmacodynamics for those with at least one EGT vs. without any EGT haplotype of the GSTZ1/MAAI gene which is located on chromosome 14q24.3.
- Total: Total of all reporting groups
Arm/Group | Lack Any EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3 | 1+ EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3 | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.0 (4.6) | 28.2 (10.4) | 26.9 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Hypothesize That Subject's Genotype Will Determine How DCA is Metabolized.
Description: Terminal half-life (the amount of time needed to clear one-half of dose of the drug).
Time Frame: 24 hours for analysis on Day 5, Clinical dose
Population: All completing subjects (2 withdrawals have no pharmacokinetic data on this parameter) The intent was to accrue 12 per group but the grant ended before that could be achieved. Subjects were recruited from a large pool but the two genetically defined subgroups are rare.
Measure: Median (Inter-Quartile Range); unit: Minutes
Groups:
- Lack Any EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3; 1+ EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3: Both dichloroacetate 2.5ug and 25mg per kg per day and is administered for five days. (Biologic randomization)
  Dichloroacetate 2.5.ug/kg (Environmental) and 25mg/kg (clinical) are administered daily for 5 days in all subjects. Subjects are admitted to the clinical research center for 6 nights. The first day subjects are administer 2.5ug/kg/day. Frequent blood samples are collected over a 24 hour period. On days 2, 3, and 4 the subjects receive a dose of DCA each day. On day 5 they receive a dose of DCA and pharmacokinetics are done for 24 hours then subjects are discharged.
Arm/Group | Lack Any EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3 | 1+ EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3
Number analyzed (Participants) | 5 | 7
Minutes | 1592 [727 to 1774] | 232 [126 to 310]
Statistical Analysis 1: Comparison: Lack Any EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3 vs 1+ EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3; We used a Wilcoxon test (and accompanying Kendal's Tau B) because these outcomes are outlier prone; Test type: Superiority or Other; p = 0.023, Wilcoxon (Mann-Whitney) — This is the primary outcome, and there is no adjustment; Kendall's Tau-B = 0.60, 95% CI 2-sided [0.35 to 0.85], Standard Error of Mean 0.127

2. Secondary Outcome: Terminal Half-life (the Amount of Time Needed to Clear One-half of the Dose of Drug)for Environmental Dose 2.5 ug/kg/Day.
Description: Terminal half-life (the amount of time needed to clear one-half of the dose of drug)for the environmental dose 2.5 ug/kg/day.
Time Frame: 24 hours for analysis on Day 5, Environmental dose
Population: same as Primary
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- No EGT Allele: No EGT allele
- At Least One EGT Allele: At least one EGT allele
Arm/Group | No EGT Allele | At Least One EGT Allele
Number analyzed (Participants) | 5 | 7
minutes | 65.4 [56.3 to 66.4] | 74.3 [58.9 to 90.4]
Statistical Analysis 1: Comparison: No EGT Allele vs At Least One EGT Allele; This is the same analysis as the previous, except we use the day 5 pharmacogenetics on the amount of time needed to clear one-half of dose of the drug. This is for the environmental dose. A positive (negative) Kendall's Tau is associated with the EGT allele being faster (slower) than lacking EGT in terms of metabolization of DCA; Test type: Superiority or Other; p = 0.42, Wilcoxon (Mann-Whitney); Kendall's Tau B = -0.23, 95% CI 2-sided [-0.23 to 0.69], Standard Error of Mean 0.23

ADVERSE EVENTS:
Time Frame: Adverse events were collected from 5/2008 to 2/2009
Arm/Group | Lack Any EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3 | 1+ EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/8
Other Adverse Events (participants affected / at risk) | 5/6 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lack Any EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3 (N=6) | 1+ EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3 (N=8)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Subject had developed a rash on his right arm where the Tegraderm from his IV was applied. It was determined he had an allergic reaction to the Tegraderm.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lack Any EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3 (N=6) | 1+ EGT Allele on GSTz1/MAAI Region of Chromosome 14q24.3 (N=8)
sleepiness (General disorders) | 5 (7) | 5 (5) — Eleven subjects on 25mg/kg of DCA complained of sleepiness following taking the drug
abdominal cramping and diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Subject complained of abdominal cramping and diarrhea which lasted for 2 days
Hives (Immune system disorders) | 0 (0) | 1 (1) — Subject complained of having hives. When examined by the principal investigator one hive was found on her right arm and was fading
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Subject had wheezes in his lower lobes of his lungs and stated he was spitting up yellow sputum. He had been having a cold when he entered the study
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) — Complained of constipation but subject was not dehydrated. A stool softener was order which resolved the problem
slow clearance of DCA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Following completion of the study when the results were being analyzed it showed that subject did not clear DCA as rapidly as other subject. It was attributed to his genotype.
headache (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject complained of a headache. It was resolved after she took a nap

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No